CLINICAL TRIAL: NCT07400614
Title: Evaluating the Impact of Energy Drink Formulas on Alertness for an Extended Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2514
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alertness
Keywords: alertness; energy; caffeine; beverage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo beverage (Placebo Comparator): Base carbonated beverage with no caffeine, taurine, or vitamins
  Interventions: Other: Flavored carbonated beverage, color-matched
- Caffeine 120 mg beverage 1 (Experimental): Carbonated beverage with varying levels of taurine and B vitamins
  Interventions: Other: All beverages are flavor and color matched
- Caffeine 120 mg beverage 2 (Experimental): Carbonated beverage with varying levels of taurine and B vitamins
  Interventions: Other: All beverages are flavor and color matched
- Caffeine 120 mg beverage 3 (Experimental): Carbonated beverage with varying levels of taurine and B vitamins
  Interventions: Other: All beverages are flavor and color matched

INTERVENTIONS:
Other: All beverages are flavor and color matched — Caffeine with varying amounts of taurine and B vitamins
  Arms: Caffeine 120 mg beverage 1; Caffeine 120 mg beverage 2; Caffeine 120 mg beverage 3
Other: Flavored carbonated beverage, color-matched — Base with 0 mg caffeine, taurine, vitamins
  Arms: Placebo beverage

SUMMARY:
The primary purpose of the research is to evaluate in healthy adults the time course effects of energy drink formulas containing 120 mg caffeine with varying levels of taurine and b vitamins on subjective alertness in the presence of cognitive load assessed hourly up to 5 hours post dose

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged 18-49 years, inclusive
* Participants self-report that they are in good health
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial
* Willing to abstain from consumption of caffeine for 12 h prior to testing
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits
* Willing to refrain from 'over the counter' medications (e.g. pain medication) and stimulant medication for 12 hours, seasonal allergy/hayfever nasal antihistamine medications for 24 hours and oral antihistamines for 48 hours prior to all test visits
* Regular caffeine consumer (at least one caffeinated beverage per day, not less than 35 mg)
* Are fluent in English (equivalent to IELTS Level 6)
* Understand the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study Investigator

Exclusion Criteria:

* Fail to meet any one of the inclusion criteria
* Currently use of prescription medication, including contraceptives
* Report hypersensitivity to caffeine
* Have experienced major trauma or major surgical event within 6 months of screening
* Have extreme dietary habits, as judged by the Investigator (high fat, very high protein diets, intermittent fasting, etc.)
* Have a history of cancer in the prior two years, except for non-melanoma skin cancer
* Have a visual impairment that cannot be corrected with glasses or contact lenses
* Have food allergies/intolerances/sensitivities to any ingredients in the study products (including coffee or related foods/beverages/products)
* Self-report excessive leisure time physical activity (> 7 strenuous bouts per week)
* Have current or chronic gastrointestinal, sleep, or psychiatric disorders
* Work night shifts or follow a variable work pattern that results in irregular sleep pattern
* Are pregnant, trying to get pregnant or lactating
* Smoke tobacco, vape nicotine or use nicotine replacement products
* Use illegal/recreational drugs
* Are unable to demonstrate adequate minimal performance on lab, computer-based cognitive tasks
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2 (unless waist to hip ratio is less than or equal to 0.85 (female) or 0.90 (male))
* Have been diagnosed with a neurological condition, or assessed as having a learning/behavioural or neurodevelopmental difference (e.g. dyslexia, autism, ADHD)
* Consume excessive caffeine intake (>400 mg per day)
* Have taken any dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffer from frequent migraines that require medication (more than or equal to 1 per month)
* Have any known active infections
* Do not have a bank account (required for payment)
* Have participated in another clinical trial within past 30 days and/or participation in another PepsiCo trial in the past 6 months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Caffeine Research Visual Analog Scale (VAS) subjective alertness factor | Change from baseline Time 0 to 240 minutes post-dose
  Created by combining 'alert' and 'tired' (reversed) responses assessed by the Caffeine Research VAS (Visual Analog Scale) adapted from Rogers et al. Subjective ratings by placing an 'x' on a line representing 0-100% to match their current state (alert, tired)

SECONDARY OUTCOMES:
Caffeine Research VAS measures (Visual Analog Scale) | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose
  Change in subjective tension factor, created by combining 'relaxed' (reversed) and 'tense' responses. Subjective ratings by placing an 'x' on a line representing 0-100% to match their current state (relaxed, tense)
Simple reaction time | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as reaction time (in milliseconds), with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Digit vigilance accuracy | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as a percentage, with a higher score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Digit vigilance reaction time | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as reaction time (in milliseconds), with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Digit vigilance false alarms | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as number of errors, with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Choice reaction accuracy (%) | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as a percentage, with a higher score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Choice reaction accuracy (milliseconds) | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as reaction time (in milliseconds), with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Rapid visual information processing accuracy | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as a percentage, with a higher score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Rapid visual information processing reaction time | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as reaction time (in milliseconds), with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)
Rapid visual information processing false alarms | Change from baseline Time 0 to 60, 120, 180, 240 & 300 minutes post-dose. Each test has duration ~21 minutes )
  Cognitive function - attention measured as number of errors, with a lower score indicating better performance using the Computerised Mental Performance Assessment System (COMPASS)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, PhD, Principal Investigator — Northumbria U Newcastle, UK
Locations (1):
- Northumbria U, Newcastle, Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No